CLINICAL TRIAL: NCT05896384
Title: A Non-randomised, Open-label Phase I Trial to Evaluate the Effect of BI 456906 at Different Dose Levels of Multiple Subcutaneous Doses in a Titration Scheme on the Single Dose Pharmacokinetics of a Combination of Ethinylestradiol and Levonorgestrel in Otherwise Healthy Women With Overweight/Obesity
Brief Title: A Study in Women With Overweight or Obesity to Test Whether Different Doses of BI 456906 Influence the Amount of a Contraceptive in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1404-0014; 2022-503146-53-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2023-06-01; First posted 2023-06-09 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Healthy
MeSH Terms: interventions — BI 456906; ethinyl estradiol, levonorgestrel drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Microgynon® (Reference treatment (R)) followed by BI 456906 and Microgynon® (Test treatment (T)) (Experimental)
  Interventions: Drug: BI 456906; Drug: Microgynon®

INTERVENTIONS:
Drug: BI 456906 — BI 456906
  Other Names: survodutide
Drug: Microgynon® — Ethinylestradiol (EE) and Levonorgestrel (LNG)

SUMMARY:
This study is open to women with overweight or obesity who are otherwise healthy. Women with a body mass index (BMI) from 27 to 40 kg/m2 can participate. The purpose of this study is to find out whether taking multiple doses of BI 456906 influences the amount of ethinylestradiol and levonorgestrel in the blood. Ethinylestradiol and levonorgestrel are ingredients of the contraceptive Microgynon®.

The study has 2 treatment periods. In Period 1, participants get 1 tablet of Microgynon®. In Period 2, participants get weekly injections of BI 456906 for 7 months. The doses of BI 456906 increase each month. At 8 specific timepoints during Period 2, participants also get 1 tablet of Microgynon®.

Participants visit the study site up to 40 times. At 8 visits, participants take Microgynon® and stay overnight at the site. During the visits, the doctors collect information about participants' health and take blood samples from the participants. They compare the amount of ethinylestradiol and levonorgestrel in the blood in Period 2 with the amounts in Period 1. Doctors also regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion Criteria:

1. Otherwise healthy women according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
2. Age of 18 to 60 years (inclusive)
3. Body mass index (BMI) of 27.0 to 40.0 kg/m2 (inclusive)
4. Signed and dated written informed consent in accordance with International Council for Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial, i.e. prior to starting any screening procedures
5. Subject fulfills any of the following criteria at least 4 weeks prior to allocation of subject number (i.e. prior to Day 1 of period 1):

   1. Use of non-hormone releasing intrauterine device (IUD) and male partner must be vasectomised (provided that partner is the sole sexual partner of the trial participant) with documented absence of sperm or use a condom
   2. Bilateral tubal ligation and male partner must be vasectomised (provided that partner is the sole sexual partner of the trial participant) with documented absence of sperm or use a condom
   3. Sexually abstinent (i.e. subjects must abstain from male-female sex)
   4. Surgically sterilised (including hysterectomy, bilateral salpingectomy, bilateral oophorectomy)
   5. Postmenopausal, defined as no menses for 1 year without an alternative medical cause (in questionable cases a blood sample with levels of follicle stimulating hormone (FSH) above 40 U/L and estradiol below 30 ng/L is confirmatory)

Exclusion Criteria:

1. Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
2. Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimetre of mercury (mmHg), diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 beats per minute (bpm)
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance and/or liver enzymes (alanine transaminase (ALT), aspartate aminotransferase (AST), gamma-glutamyl transpeptidase (GGT)) and/or pancreatic enzymes (amylase lipase) above upper limit of normal range +10% at screening examination, confirmed by a repeat test
4. Any evidence of a concomitant disease assessed as clinically relevant by the investigator
5. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
6. History of either chronic or acute pancreatitis
7. Cholecystectomy, and/or prior surgery of the gastrointestinal (GI) tract (including bariatric surgery) or any relevant anatomical malformation of the GI tract that could interfere with the pharmacokinetics of the trial medication (investigational medicinal product (IMP) or auxiliary medicinal product (AxMP)) - except appendectomy or simple hernia repair
8. Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
9. History of relevant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2023-12-21 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2025-03-26 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of ethinylestradiol in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) | up to Week 29
Maximum measured concentration of ethinylestradiol in plasma (Cmax) | up to Week 29
Area under the concentration-time curve of levonorgestrel in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) | up to Week 29
Maximum measured concentration of levonorgestrel in plasma (Cmax) | up to Week 29

CONTACTS AND LOCATIONS:
Locations (1):
- Charité Research Organisation GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com